CLINICAL TRIAL: NCT05183477
Title: Fast Track in the Emergency Department for Wrist and Scaphoid Fractures: a Randomised Trial
Brief Title: Fast Track for Wrist and Scaphoid Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator's departure
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-02140
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Wrist Fracture; Scaphoid Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fast track (Experimental): patients arriving at Emergency Department with suspected wrist or scaphoid fracture, randomly allocated to the fast track pathway (xray requested at triage by nurse)
  Interventions: Other: fast track
- normal pathway (Active Comparator): patients arriving at Emergency Department with suspected wrist or scaphoid fracture, randomly allocated to waiting room and than medical examination before asking for xrays
  Interventions: Other: normal pathway

INTERVENTIONS:
Other: fast track — short cut for the request of xrays directly at triage
  Arms: fast track
Other: normal pathway — x-ray would be required according to doctor's clinical evaluation.
  Arms: normal pathway

SUMMARY:
This is a mono centric, prospective, randomised trial on the implementation and assessment of a shortened pathway for mono-trauma of the wrist and suspected fracture of distal radius and/or ulna and/or scaphoid bone.

DETAILED DESCRIPTION:
Patients will be randomised into two groups: fast track and normal pathway. At the arrival in the Emergency Department a triage will be performed. In case of met inclusion criteria the patient will sign the informed consent and will be randomised in one of the two study groups.

The fast track group will be straightforwardly evaluated for absence of exclusion criteria (in case of exclusion criteria present the investigators will follow the normal pathway and the patient will not be included in the study). Then, patients will be assessed with an ad hoc checklist and then sent for x-ray performance, if necessary. After the x-ray the patients will be examined by an emergency physician that will have the opportunity to request new x-ray views if necessary.

The normal pathway group will go straight to medical examination as soon as possible, depending on waiting times in the Emergency Department.

Investigators will collect anagraphical data, waiting times, time to x-ray, overall length of stay in the Emergency Department, patients' and staff's satisfaction for the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adults patients presenting at the emergency dept with suspected scaphoid or wrist fracture
* monotrauma
* written informed consent

Exclusion Criteria:

* patients younger than 18 yr
* pregnant women
* either vascular or neural impairment
* signs of open fracture
* multiple trauma patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
number of x rays requested | From admission to discharge, up to 2.5 hours
  the number of xray requested

SECONDARY OUTCOMES:
waiting time before examination | From admission to discharge, up to 2.5 hours
waiting time before xray | From admission to discharge, up to 2.5 hours
total length of stay in the emergency department | From admission to discharge, up to 2.5 hours
patient's satisfaction | From admission to discharge, up to 2.5 hours
  Patients' satisfaction will be tested with the help of the brief emergency department patient satisfaction scale (BEPSS). The questionnaire consists of 20 questions and for each item, a response scale form 1 (completely disagree) to 4 (completely agree) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Uccella, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ospedale Regionale di Lugano - ORL, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
no plan at the moment

REFERENCES:
- [Background] Mallee WH, Walenkamp MMJ, Mulders MAM, Goslings JC, Schep NWL. Detecting scaphoid fractures in wrist injury: a clinical decision rule. Arch Orthop Trauma Surg. 2020 Apr;140(4):575-581. doi: 10.1007/s00402-020-03383-w. Epub 2020 Mar 3. PMID 32125528
- [Background] Walenkamp MM, Bentohami A, Slaar A, Beerekamp MS, Maas M, Jager LC, Sosef NL, van Velde R, Ultee JM, Steyerberg EW, Goslings JC, Schep NW. The Amsterdam wrist rules: the multicenter prospective derivation and external validation of a clinical decision rule for the use of radiography in acute wrist trauma. BMC Musculoskelet Disord. 2015 Dec 18;16:389. doi: 10.1186/s12891-015-0829-2. PMID 26682537
- [Background] Chudleigh J. Nurse requested X-rays in A&E department. Emerg Nurse. 2004 Feb;11(9):32-6. doi: 10.7748/en2004.02.11.9.32.c1146. No abstract available. PMID 15000019
- [Background] Streppa J, Schneidman V, Biron AD. Requesting wrist radiographs in emergency department triage: developing a training program and diagnostic algorithm. Adv Emerg Nurs J. 2014 Jan-Mar;36(1):62-77. doi: 10.1097/TME.0000000000000005. PMID 24487265
- [Background] van den Brand CL, van Leerdam RH, van Ufford JH, Rhemrev SJ. Is there a need for a clinical decision rule in blunt wrist trauma? Injury. 2013 Nov;44(11):1615-9. doi: 10.1016/j.injury.2013.07.006. Epub 2013 Jul 31. PMID 23915492